CLINICAL TRIAL: NCT02825095
Title: Management of Malignant Pleural Effusion - Indwelling Pleural Catheter or Talc Pleurodesis ; a Prospective Randomized Controlled Study.
Brief Title: Management of Malignant Pleural Effusion - Indwelling Pleural Catheter or Talc Pleurodesis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0371-15rmb
Record Dates: First submitted 2016-04-04; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Pleural Effusion, Malignant; Lung Neoplasms
Keywords: malignant pleural effusion,talc pleurodesis,quality of life
MeSH Terms: conditions — Pleural Effusion, Malignant; Lung Neoplasms | interventions — Anesthesia, Local; Lidocaine; Chest Tubes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Talc Pleurodesis (Active Comparator): For patients in this group, chest tube type PIGTAIL 10 - 14 Fr will be inserted by by chest ultrasound guided and under local anesthesia, allowing good draining of the hemithorax, in case of fluid discharges less than 250 cc/24, talc pleurodesis will be performed, chest tube will be removed 24 - 48 hours later on. the patient will be admitted in the hospital during the whole procedure course.
  If the patient developed non expanded - trapped lung post chest tube insertion, or if he had persistence high chest tube output for more than 10 days, then the patient will remain with the PIGTAIL as an Indwelling Pleural Catheter.
  Interventions: Procedure: Talc Pleurodesis; Procedure: chest ultrasound; Drug: Local anesthesia; Procedure: Chest Tube
- Indwelling Pleural Catheter (Active Comparator): All patients from this group will have Indwelling Pleural Catheter insertion type PLEURAX inserted by ultrasound guided and under local anesthesia.
  the patient and his/her family will be instructed and educated about the proper way of using the catheter, and how to perform pleural draining at home.
  the duration of treatment with the Pleurax depends on the rate and amount of pleural effusion draining.
  Interventions: Procedure: Indwelling Pleural Catheter; Procedure: chest ultrasound; Drug: Local anesthesia

INTERVENTIONS:
Procedure: Talc Pleurodesis — chest tube type PIGTAIL 10 - 14 Fr will be inserted to the pleural space. In case of fluid discharges less than 250 cc/24, talc pleurodesis will be performed
  Arms: Talc Pleurodesis
Procedure: Indwelling Pleural Catheter — Indwelling Pleural Catheter type PLEURAX will be inserted to the pleural space. the patients will be discharged with the pleural catheter.
  Arms: Indwelling Pleural Catheter
Procedure: chest ultrasound — All insertion of a chest drain will be guided by ultrasound
Drug: Local anesthesia — Inserting a chest drain will be after local anesthesia with 10-20 mL of Lidocaine hydrochloride 20MG/ML - Esracain injection 2%
  Other Names: Lidocaine hydrochloride; Esracain injection 2%
Procedure: Chest Tube — chest tube type PIGTAIL 10 - 14 Fr will be inserted to the pleural space. In case of fluid discharges less than 250 cc/24, talc pleurodesis will be performed
  Other Names: PIGTAIL
  Arms: Talc Pleurodesis

SUMMARY:
Prospective study of the effect of Talc Pleurodesis vs. Indwelling Pleural catheter in treatment of patients with malignant pleural effusion

DETAILED DESCRIPTION:
Randomized prospective study that will include 120 patients with malignant pleural effusion with high rate of accumulation; less than one month, The patients will be divided randomly for two groups, each group 60 patients, the first group will undergoes talc pleurodesis, the second group will undergoes Indwelling Pleural catheter insertion.

The two groups will be followed up for one year, starting at the time of intervention, after 14 days of intervention, after 30 days of intervention, once monthly for one year.

The patients will be evaluated according to the rate of complication; need for further intervention in each group, improvement of the quality of life, respiratory improvement, radiological evaluation based on chest Xray findings, rate and duration of admissions that are related to pleural effusion during the year of study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent symptomatic pleural effusion, the diagnosis was obtained by : - positive cytology for malignant cells in the fluid.

   * patients well known for malignancy, with exudative pleural effusion with no alternative diagnosis.
   * pleural biopsy - surgically obtained - with diagnosis of pleural malignancy
   * microscopic intraoperative findings suggestive of pleural malignancy.
2. Patients who underwent prior to involvement in the study, draining of the pleural fluid with symptomatic improvement.
3. Patients with rate of fluid accumulation less than 30 days.
4. Patient who signed informed consent about being involved in the study.

Exclusion Criteria:

1. Patients under the age of 18 years.
2. Female patients who are Pregnant or nursing.
3. Patients with rate of pleural effusion accumulation is more than 30 days.
4. Patients who didn't show clinical improvement post proper draining of the fluid
5. Patients who are hemodynamically or respiratory unstable.
6. Patients with Empyema.
7. Patients who are non functioning/ not active according to the Performance status.
8. The type of malignancy which cause the malignant pleural effusion is Lymphoma.
9. Patient who underwent pneumonectomy at the side of the fluid.
10. previous pleurodesis at the side of pleural effusion.
11. Chylothorax in the initial pleural tapping.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
change in Quality of Life | one year of regular follow up.
  the patients will be followed up 14 days post intervention, 30 days, once monthly for 12 months, the patient will fill questioner every month evaluating the quality of life, the daily activities and the degree of shortness of breath.

SECONDARY OUTCOMES:
procedure and admissions | one year
  The patients will be evaluated for the number of admissions: e.g: how many times he/she was admitted to the hospital, duration of admissions; how many days he was admitted in the hospital each time and procedure related to pleural effusion; types and number of procedures

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Heffner JE, Klein JS. Recent advances in the diagnosis and management of malignant pleural effusions. Mayo Clin Proc. 2008 Feb;83(2):235-50. doi: 10.4065/83.2.235. PMID 18241636
- [Background] Roberts ME, Neville E, Berrisford RG, Antunes G, Ali NJ; BTS Pleural Disease Guideline Group. Management of a malignant pleural effusion: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii32-40. doi: 10.1136/thx.2010.136994. No abstract available. PMID 20696691
- [Background] Sahn SA. Pleural diseases related to metastatic malignancies. Eur Respir J. 1997 Aug;10(8):1907-13. doi: 10.1183/09031936.97.10081907. PMID 9272937
- [Background] Uzbeck MH, Almeida FA, Sarkiss MG, Morice RC, Jimenez CA, Eapen GA, Kennedy MP. Management of malignant pleural effusions. Adv Ther. 2010 Jun;27(6):334-47. doi: 10.1007/S12325-010-0031-8. Epub 2010 Jun 10. PMID 20544327
- [Background] Chernow B, Sahn SA. Carcinomatous involvement of the pleura: an analysis of 96 patients. Am J Med. 1977 Nov;63(5):695-702. doi: 10.1016/0002-9343(77)90154-1. No abstract available. PMID 930945
- [Background] American Thoracic Society. Management of malignant pleural effusions. Am J Respir Crit Care Med. 2000 Nov;162(5):1987-2001. doi: 10.1164/ajrccm.162.5.ats8-00. No abstract available. PMID 11069845
- [Background] Nam HS. Malignant pleural effusion: medical approaches for diagnosis and management. Tuberc Respir Dis (Seoul). 2014 May;76(5):211-7. doi: 10.4046/trd.2014.76.5.211. Epub 2014 May 29. PMID 24920947
- [Background] Zarogoulidis K, Zarogoulidis P, Darwiche K, Tsakiridis K, Machairiotis N, Kougioumtzi I, Courcoutsakis N, Terzi E, Zaric B, Huang H, Freitag L, Spyratos D. Malignant pleural effusion and algorithm management. J Thorac Dis. 2013 Sep;5 Suppl 4(Suppl 4):S413-9. doi: 10.3978/j.issn.2072-1439.2013.09.04. PMID 24102015
- [Background] Olden AM, Holloway R. Treatment of malignant pleural effusion: PleuRx catheter or talc pleurodesis? A cost-effectiveness analysis. J Palliat Med. 2010 Jan;13(1):59-65. doi: 10.1089/jpm.2009.0220. PMID 19839739
- [Background] Chee A, Tremblay A. The use of tunneled pleural catheters in the treatment of pleural effusions. Curr Opin Pulm Med. 2011 Jul;17(4):237-41. doi: 10.1097/MCP.0b013e3283463dac. PMID 21460729
- [Background] Srour N, Amjadi K, Forster A, Aaron S. Management of malignant pleural effusions with indwelling pleural catheters or talc pleurodesis. Can Respir J. 2013 Mar-Apr;20(2):106-10. doi: 10.1155/2013/842768. PMID 23616967